CLINICAL TRIAL: NCT05141903
Title: Dietary Study of a Complex Oligosaccharide With and Without a Probiotic Following Antibiotic Treatment in Healthy Volunteers
Brief Title: Dietary Supplement With and Without a Probiotic and/or Antibiotic
Status: Completed | Type: Observational
Sponsor: Prolacta Bioscience (Industry)
Responsible Party: Sponsor
Other Study IDs: 21-CT-003
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Anti-Bacterial Agents; Probiotics; Dietary Supplements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Urine, and Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Arm 1: D1-D5: Antibiotics (3x daily)
  Interventions: Dietary Supplement: Antibiotic
- Arm 2: D1-D5: Antibiotics (3x daily) D1-D14: Probiotic D1-D28: 18 g HMO concentrate (9g twice daily)
  Interventions: Dietary Supplement: Antibiotic; Dietary Supplement: HMO Concentrate; Dietary Supplement: Probiotic
- Arm 3: D1-D5: Antibiotics (3x daily) D1-D14: Probiotic
  Interventions: Dietary Supplement: Antibiotic; Dietary Supplement: Probiotic
- Arm 4: D1-D5: Antibiotics (3x daily) D1-D14: Probiotic + 18 g HMO concentrate (9g twice daily) D15-D28: 22g Food Supplement (11 g daily)
  Interventions: Dietary Supplement: Antibiotic; Dietary Supplement: HMO Concentrate; Dietary Supplement: Probiotic; Dietary Supplement: Food Supplement
- Arm 5: D1-D5: Antibiotics (3x daily) D1-D14: Probiotic D1-D28: 22g Food Supplement (11 g daily)
  Interventions: Dietary Supplement: Antibiotic; Dietary Supplement: Probiotic; Dietary Supplement: Food Supplement

INTERVENTIONS:
Dietary Supplement: Antibiotic — Vancomycin (250 mg/dose), Metronidazole (500 mg/dose)
Dietary Supplement: HMO Concentrate — Concentrated milk fortifiers from donor human milk
  Groups: Arm 2; Arm 4
Dietary Supplement: Probiotic — B. infantis
  Groups: Arm 2; Arm 3; Arm 4; Arm 5
Dietary Supplement: Food Supplement — Synthetic powder containing 2'-fucosyllactose (2'-FL) and lactoneotetraose (LNnT)
  Groups: Arm 4; Arm 5

SUMMARY:
Complex oligosaccharides can alter the gut microbiome by aiding in the growth of certain organisms, and possibly, inhibiting others. The synergy with a probiotic may enhance gastrointestinal colonization.

DETAILED DESCRIPTION:
The study will evaluate the synergy of the use of a complex oligosaccharide with and without a probiotic on the human microbiome in healthy volunteers who have received antibiotics. The combination should support general gastrointestinal health.

This study is a multi-dose randomized cohort trial using 18 subjects per cohort for a total of 90 healthy adult volunteers ages 18-75.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between the ages of 18-75 years (subjects must be 18-75 at the time of consent) who can provide proof of vaccination against SARS-CoV-2. Proof may be a physical or electronic record of vaccination or self-attestation (to include approximate vaccination date and manufacturer of vaccine) if a copy of the vaccination record is not available
* Subjects must have a BMI of 18 - 30 at screening visit
* Willingness to complete study specific questionnaires
* Willingness to complete journal to record IP dosing times, Bristol stool scores, and IP flavor questionnaires
* Willingness to complete all study procedures, clinic visits, and provide required biospecimen samples
* Willingness to collect and process stool samples at home and transport stool samples to clinic
* Sexually active females of child-bearing potential must agree to use highly effective methods of contraception during heterosexual intercourse throughout the study period and for three days following discontinuation of IP, whichever comes later. Examples of highly effective methods include the use of two forms of contraception with one being an effective barrier method (e.g., a condom and spermicide used together), or have a vasectomised partner. Abstinence is acceptable as a life-style choice. Female subjects who utilize hormonal contraceptives as one of their birth control methods must have used the same method for at least 3 months before study dosing
* Provide informed consent

Exclusion Criteria:

* Subjects with a BMI of 17 or less or 31 or greater are excluded
* Women who are pregnant or breastfeeding, or intend to become pregnant during the course of this study
* Subjects who intend to take a probiotic during the study
* Subjects with self-reported diarrhea on day 1 prior to dosing, whereby diarrhea is defined as two or more episodes of watery and/or unformed stool within 24 hours
* Alcohol or drug abuse during the last 12 months, including passing a screen for drugs of abuse at screening and day 1 of the study
* Unstable medical condition, in the opinion of the investigator
* Subject with a history of allergy to the study antibiotics
* Clinically significant abnormal laboratory test results at screening
* Subjects who are unable or unwilling to provide stool samples on a regular basis as per study protocol
* Participation in a clinical research trial within 30 days prior to screening
* Unable to give informed consent
* Any condition which may preclude subject's ability to comply with and complete the study or may pose a risk to the health of the subject
* Known carriers of C. difficile prior to study start, as determined by qPCR of stool
* Known carriers of vancomycin-resistant enterococci (VRE) prior to study start, as determined by stool culture
* Subjects with history of lactose intolerance

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy Adults, ages 18-75.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-06-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences, Cypress, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Antibiotics Alone: Antibiotics (Only)
- Antibiotics, Probiotic, HMO: Antibiotics, Probiotic, HMO Concentrate
- Antibiotics Probiotic: Antibiotics, Probiotic
- Antibiotics, Probiotic, HMO, Food: Antibiotics, Probiotic, HMO concentrate, Food Supplement
- Antibiotics, Probiotic, Food: Antibiotics, Probiotic, Food Supplement
Period: Overall Study
Arm/Group | Antibiotics Alone | Antibiotics, Probiotic, HMO | Antibiotics Probiotic | Antibiotics, Probiotic, HMO, Food | Antibiotics, Probiotic, Food
Started | 19 | 19 | 18 | 18 | 18
Completed | 18 | 17 | 17 | 18 | 18
Not Completed | 1 | 2 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0
Not completed — Other | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Antibiotics Alone: D1-D5: Antibiotics (3x daily)
  Antibiotic: Vancomycin (250 mg/dose), Metronidazole (500 mg/dose)
- Antibiotics, Probiotic, HMO: D1-D5: Antibiotics (3x daily) D1-D14: Probiotic D1-D28: 18 g HMO concentrate (9g twice daily)
  Antibiotic: Vancomycin (250 mg/dose), Metronidazole (500 mg/dose)
  HMO Concentrate: Concentrated milk fortifiers from donor human milk
  Probiotic: B. infantis
- Antibiotics, Probiotic: D1-D5: Antibiotics (3x daily) D1-D14: Probiotic
  Antibiotic: Vancomycin (250 mg/dose), Metronidazole (500 mg/dose)
  Probiotic: B. infantis
- Antibiotics, Probiotic, HMO, Food: D1-D5: Antibiotics (3x daily) D1-D14: Probiotic + 18 g HMO concentrate (9g twice daily) D15-D28: 22g Food Supplement (11 g daily)
  Antibiotic: Vancomycin (250 mg/dose), Metronidazole (500 mg/dose)
  HMO Concentrate: Concentrated milk fortifiers from donor human milk
  Probiotic: B. infantis
  Food Supplement: Synthetic powder containing 2'-fucosyllactose (2'-FL) and lactoneotetraose (LNnT)
- Antibiotics, Probiotic, Food: D1-D5: Antibiotics (3x daily) D1-D14: Probiotic D1-D28: 22g Food Supplement (11 g daily)
  Antibiotic: Vancomycin (250 mg/dose), Metronidazole (500 mg/dose)
  Probiotic: B. infantis
  Food Supplement: Synthetic powder containing 2'-fucosyllactose (2'-FL) and lactoneotetraose (LNnT)
- Total: Total of all reporting groups
Arm/Group | Antibiotics Alone | Antibiotics, Probiotic, HMO | Antibiotics, Probiotic | Antibiotics, Probiotic, HMO, Food | Antibiotics, Probiotic, Food | Total
Number analyzed (Participants) | 19 | 19 | 18 | 18 | 18 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 1 | 1
  Between 18 and 65 years | 14 | 18 | 14 | 16 | 16 | 78
  >=65 years | 5 | 1 | 4 | 2 | 1 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 7 | 7 | 10 | 42
  Male | 7 | 13 | 11 | 11 | 8 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 5 | 5 | 4 | 24
  Not Hispanic or Latino | 14 | 14 | 13 | 13 | 14 | 68
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 4 | 5 | 7 | 3 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 3 | 0 | 2 | 10
  White | 13 | 11 | 10 | 10 | 11 | 55
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 0 | 0 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 18 | 18 | 18 | 92
Baseline Levels of B. Infantis [Mean (Standard Deviation); unit: copies/ng DNA] | 27.00 (0.00) | 31.25 (82.27) | 27.00 (0.00) | 27.00 (0.00) | 27.00 (0.00) | 27.8 (36.2)

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Changes in Microbiome Species Abundance and Diversity From Baseline Until End of Study (Day 35)
Description: Evaluation of HMO supporting gut colonization of B.infantis in healthy adult volunteers with microbiome disruption by antibiotics. Stool samples were taken from subjects at regular intervals and prepared for DNA extraction and microbiome analysis. Following DNA extraction, samples were analyzed using subspecies-specific qPCR analysis to evaluate B.infantis colonization and monitor overall shifts using primers that target universal 16S rRNA gene shared by bacteria by log-fold changes.
Time Frame: Baseline, Day, 5, 14, 35
Population: All participants assigned to an arm and were able to provide adequate evaluable samples for DNA analysis
Measure: Geometric Mean (Standard Deviation); unit: copies/ng DNA
Groups:
- Antibiotics, Probiotics, HMO: Antibiotics, Probiotic, HMO Concentrate
- Antibiotics Probiotics: Antibiotics and Probiotic
- Antibiotics, Probiotics, HMO, Food: Antibiotics, Probiotic, HMO concentrate, Food Supplement
- Antibiotics, Probiotics, Food: Antibiotics, Probiotic, Food Supplement
Arm/Group | Antibiotics Alone | Antibiotics, Probiotics, HMO | Antibiotics Probiotics | Antibiotics, Probiotics, HMO, Food | Antibiotics, Probiotics, Food
Number analyzed (Participants) | 19 | 17 | 17 | 18 | 18
copies/ng DNA
  Baseline | 27.00 (0.00) | 31.25 (82.27) | 27.00 (0.00) | 27.00 (0.00) | 27.00 (0.00)
  Day 5 | 27.00 (0.00) | 383.41 (862.67) | 535.35 (708.21) | 204.11 (312.05) | 431.26 (883.43)
  Day 14 | 28.08 (6.87) | 26877.59 (69845.62) | 1868.09 (10150.73) | 21736.64 (50622.14) | 45466.96 (81975.89)
  Day 35 | 27.00 (0.00) | 311.22 (14917.81) | 77.15 (1857.25) | 88.78 (1249.73) | 170.03 (5638.54)
Statistical Analysis 1: Comparison: Antibiotics Alone vs Antibiotics, Probiotics, HMO; Dose Group 2 B. infantis levels compared to control group (antibiotic only) with changes over time; Test type: Superiority; p < 0.0001, Mixed Models Analysis — (Dose group * Time); Dfn, Dfd = 11, 369 F Value = 24.31
Statistical Analysis 2: Comparison: Antibiotics Alone vs Antibiotics Probiotics; Dose Group 3 B. infantis levels compared to control group (antibiotic only) with changes over time; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Dose group * Time; Dfn, Dfd = 11, 370 F value = 14.87
Statistical Analysis 3: Comparison: Antibiotics, Probiotics, HMO vs Antibiotics Probiotics; Dose Group 2 (with HMO) B. infantis levels compared to dose Group 3 (without HMO) with changes over time; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Dose Group * Time; Dfn, Dfd = 11, 351 F value = 8.606

2. Secondary Outcome: Changes in Immune Markers Assessment at Day 5, 14 and 28
Description: Blood samples were collected at regular intervals for serum immunological parameters (LAP-TGFB, MCP1, MIP-1) to assess metabolite levels.
Time Frame: Baseline-28 days
Population: Analysis of Group 1 control vs Group 2 +HMO to assess impact of study product. Subjects who provided evaluable samples for all time points were evaluated for clinical pharmacology endpoints. DATA WERE COLLECTED FOR ONLY GROUPS 1 AND 2.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Antibiotics Alone | Antibiotics, Probiotic, HMO
Number analyzed (Participants) | 19 | 17
ng/mL
  LAP-TGFB - baseline | 34.3 (8.1) | 37.6 (9.6)
  LAP-TGFB - Day 5 | 34.3 (7.7) | 34.6 (7.8)
  LAP-TGFB - Day 14 | 29.7 (9.0) | 34.7 (8.1)
  LAP-TGFB - Day 28 | 30.2 (9.3) | 32.9 (5.9)
  MCP1 - Baseline | 405.6 (211.3) | 399.7 (253.3)
  MCP1 - Day 5 | 416.6 (214.0) | 401.8 (215.5)
  MCP1 - Day 14 | 476.8 (243.8) | 411.1 (199.1)
  MCP1 - Day 28 | 464.3 (250.6) | 433.8 (187.3)
  MIP - Baseline | 385.7 (106.9) | 358.2 (228.7)
  MIP - Day 5 | 429 (129.9) | 391.9 (231.0)
  MIP - Day 14 | 383.6 (226.1) | 361.6 (224.2)
  MIP - Day 28 | 315.1 (134.5) | 322.0 (226.7)

3. Secondary Outcome: Blood Pressures of Subjects From Baseline to Day 35
Description: Clinical assessments from baseline throughout study to assess vital signs of subject safety (blood pressure [BP]). Descriptive statistics performed by dose group and visit.
Time Frame: Day 0 - 35
Population: All participants assigned to an arm and were able to provide blood pressure data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Antibiotics Alone | Antibiotics, Probiotic, HMO | Antibiotics Probiotic | Antibiotics, Probiotic, HMO, Food | Antibiotics, Probiotic, Food
Number analyzed (Participants) | 19 | 19 | 18 | 18 | 18
mmHg
  Systolic Blood Pressure (mmHg) - Baseline | 123 (13.8) | 125 (19) | 127 (15.2) | 117 (11) | 121 (15.6)
  Systolic Blood Pressure (mmHg) - Day 35 | 128 (16.6) | 127 (17.3) | 130 (18.7) | 121 (14.8) | 120 (18.1)
  Diastolic Blood Pressure (mmHg) - Baseline | 75 (5.6) | 77 (11.7) | 76 (9.7) | 71 (8.5) | 73 (7.9)
  Diastolic Blood Pressure (mmHg) - Day 35 | 75 (7.4) | 74 (10) | 77 (12.1) | 73 (10) | 71 (10.3)

4. Secondary Outcome: Heart Rates of Subjects From Baseline to Day 35
Description: Clinical assessment from baseline throughout study to assess vital signs of subject safety (heart rate). Descriptive statistics performed by dose group and visit.
Time Frame: Day 0-35
Population: All participants assigned to an arm and were able to provide heart rate data.
Measure: Mean (Standard Deviation); unit: beats per minute
Groups:
- Antibiotic, Probiotic: Antibiotics, probiotic
Arm/Group | Antibiotics Alone | Antibiotics, Probiotic, HMO | Antibiotic, Probiotic | Antibiotics, Probiotic, HMO, Food | Antibiotics, Probiotic, Food
Number analyzed (Participants) | 19 | 19 | 18 | 18 | 18
beats per minute
  Heart rate - Baseline | 66 (10.9) | 66 (8.7) | 68 (8.1) | 70 (11.9) | 71 (7.4)
  Heart rate - Day 35 | 69 (10.9) | 72 (16.2) | 73 (11.1) | 66 (11.9) | 68 (10.1)

5. Secondary Outcome: Respiratory Rates of Subjects From Baseline to Day 35
Description: Clinical assessment from baseline throughout study to assess vital signs of subject safety (respiratory rate). Descriptive statistics performed by dose group and visit.
Time Frame: Day 0-35
Population: All participants assigned to an arm and were able to provide respiration rates
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Antibiotics Alone | Antibiotics, Probiotic, HMO | Antibiotic, Probiotic | Antibiotics, Probiotic, HMO, Food | Antibiotics, Probiotic, Food
Number analyzed (Participants) | 19 | 19 | 18 | 18 | 18
breaths per minute
  Respirations - Baseline | 15 (1.6) | 15 (1.1) | 15 (1.2) | 15 (1.0) | 16 (1.2)
  Respirations - Day 35 | 15 (1.1) | 15 (1.4) | 15 (1.7) | 15 (1.1) | 14 (0.9)

6. Secondary Outcome: Temperatures of Subjects From Baseline to Day 35
Description: Clinical assessment from baseline throughout study to assess vital signs of subject safety (temperature).
Time Frame: Day 0-35
Population: All participants assigned to an arm and were able to provide temperatures.
Measure: Mean (Standard Deviation); unit: deg C
Arm/Group | Antibiotics Alone | Antibiotics, Probiotic, HMO | Antibiotic, Probiotic | Antibiotics, Probiotic, HMO, Food | Antibiotics, Probiotic, Food
Number analyzed (Participants) | 19 | 19 | 18 | 18 | 18
deg C
  Temperature - Baseline | 36.8 (0.21) | 36.7 (0.24) | 36.9 (0.24) | 36.8 (0.28) | 36.9 (0.22)
  Temperature - Day 35 | 36.9 (0.14) | 36.8 (0.19) | 36.8 (0.13) | 36.8 (0.28) | 36.8 (0.28)

ADVERSE EVENTS:
Time Frame: up to 7 weeks (D1 through D35)
Groups:
- Arm 1: Antibiotics (Only)
- Arm 2: Antibiotics, Probiotic, HMO Concentrate
- Arm 3: Antibiotics, Probiotic
- Arm 4: Antibiotics, Probiotic, HMO concentrate, Food Supplement
- Arm 5: Antibiotics, Probiotic, Food Supplement
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 4/19 | 4/19 | 6/18 | 7/18 | 2/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=19) | Arm 2 (N=19) | Arm 3 (N=18) | Arm 4 (N=18) | Arm 5 (N=18)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GI Hypermotility (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry Lips (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SARS-COV-2 Test Positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT05141903/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT05141903/SAP_001.pdf